CLINICAL TRIAL: NCT02272712
Title: The Effectiveness of Online Treatment for Insomnia in Cancer Survivors: A Randomized Controlled Trial
Brief Title: The Effectiveness of Online Treatment for Insomnia in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20140224-01H
Record Dates: First submitted 2014-10-06; First posted 2014-10-23 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Chronic Insomnia
Keywords: cancer survivor; computerized treatment; symptom management
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioural Therapy (Experimental): A 6-week online cognitive-behavioural treatment for insomnia. Each week focuses on a different topic consistent with the cognitive-behavioural theory of insomnia.
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Control Condition (No Intervention): The online attention matched control arm will provide education about sleep without any focus on the active ingredients that constitute the intervention group.

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — psychoeducation about insomnia, relaxation training, sleep restriction, stimulus control, hypnotic tapering under direction of a physician, cognitive therapy, sleep hygiene
  Arms: Cognitive Behavioural Therapy

SUMMARY:
Chronic insomnia affects more than 25% of cancer survivors, a rate double that of the general population. The Pan-Canadian sleep guideline for adults with cancer recommends Cognitive-Behavioral Therapy for Insomnia (CBT-I) as the best treatment. Major problems, however, are the lack of available CBT-I at cancer centers and the lack of information about possible side-effects of CBT-I. To address this issue, our study will evaluate the effectiveness and potential short-term side-effects of an online version of CBT-I. It is expected that when compared to cancer survivors who receive an online sleep education program, those who receive online CBT-I will experience improved sleep, mood, and quality of life, as well as reduced anxiety and fatigue.

DETAILED DESCRIPTION:
Insomnia is a common adverse effect of cancer and its treatment. More than 25% of cancer survivors meet diagnostic criteria, a rate at least two times higher than that of the general population. Despite the pervasiveness of the problem, insomnia is underdiagnosed and undertreated in cancer survivors, resulting in significant suffering and associated consequences such as fatigue, cognitive issues, mood disturbance, functional disability, decreased quality of life, and immunosuppression. Consistent with recent evidence that group cognitive behavioral therapy for insomnia (CBT-I) is effective in treating insomnia in cancer survivors, CBT-I is recommended as first line treatment in the new Pan-Canadian practice guideline for sleep disturbance in adults with cancer. A major barrier to practical application of this recommendation however, is the lack of appropriately trained professionals at cancer centres. Moreover, it is assumed that in contrast to pharmacotherapy, CBT-I is free of treatment-related side-effects; however, we have no knowledge of symptoms that may be experienced by cancer survivors and/or exacerbated during CBT-I treatment (e.g., increased fatigue, cognitive impairment) because such effects are not systematically monitored. With the goal of improved access to CBT-I, online versions have been developed. One initial evaluation has been conducted in cancer patients with promising results, although limitations of the study include a small sample size (n = 28), control condition that failed to match for modality and time, lack of follow-up data, and failure to investigate potential side effects during treatment. Further inquiry is clearly warranted and consistent with insights of Canadian cancer patients who have suggested the use of technology as a factor that would facilitate their participation in an insomnia treatment program.

Specific research questions to be addressed in our proposed two-group, randomized, controlled trial include: 1) Do cancer survivors with chronic insomnia who receive a 6-week, internet-based CBT-I treatment have greater improvement in insomnia severity and other secondary sleep and quality of life outcomes, than participants in an online sleep education control group? 2) Are there short-term side-effects associated with CBT-I for cancer survivors (i.e., do participants get worse before they get better)?

Adult outpatients diagnosed with any type of cancer (stages I-III), completed active treatment for at least 1 month (with the exception of hormone therapy) and without cancer recurrence will be will be recruited from The Ottawa Hospital Cancer Centre and Cancercare Manitoba (n = 150). All will meet established diagnostic and research criteria for chronic insomnia. Prior to acceptance in the study, the procedures will be fully explained, inclusion/exclusion criteria assessed, and formal consent obtained. Once accepted into the study, participants will be randomized (stratified by hormone therapy-yes or no) to one of the two study arms. Online assessment measures (insomnia severity, pre-sleep arousal, beliefs about sleep, fatigue, mood, anxiety, quality of life) will be completed at the baseline period, at week 6 (post treatment), and at 3 month follow-up; however, online diary assessments of sleep parameters and potential side-effects (fatigue, affect, cognition, pain, drug dosing) will be entered daily and potential side-effects will also be assessed online weekly through the course of treatment. Analyses will involve mixed modeling and latent growth curve models.

The computerized intervention evaluated in this study has the potential to bridge an existing gap in knowledge translation by providing cancer survivors widespread access to CBT-I in a cost-effective manner. The study will also investigate potential short-term side-effects of online CBT-I so that patients can be fully informed when making treatment decisions. The online program could serve as the foundation of a stepped care model as recommended in the Pan-Canadian sleep guideline for adults with cancer. Overall, by reducing the burden of residual effects of cancer and its treatments, this research aims to enhance quality of life for cancer survivors in Canada and elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients with a diagnosis of any type of cancer (stages I-III) as long as active treatment is complete for at least 1 month (with the exception of hormone therapy) and there is no diagnosis of cancer recurrence
* Presence of a) difficulty with initiating or maintaining sleep or early morning awakening ≥ 30 minutes, b) daytime impairment (e.g., reduced concentration, fatigue, irritability), c) persistence of problem for at least 3 months, occurring ≥ 3 nights per week, with d) adequate opportunity for sleep and e) not entirely attributable to a mental or physical health disorder, f) access to high speed internet

Exclusion Criteria:

* Diagnosis of cancer recurrence
* Presence of symptoms suggestive of acute suicidality, current mania, schizophrenia, or head injury
* Shift work
* Weekly alcohol use in excess of 14 drinks per week for males and 12 drinks per week for females
* Current or previous cognitive behavioral therapy for insomnia
* Non-residents of Ontario

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2014-05; Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (Morin & Espie, 2003) | October 2016 - October 2019, up to 3 years
  A psychometrically sound 7-item self-report measure of perceived sleep impairment. Each item is rated using a five-point Likert scale ranging from 0 (not at all) to 4 (very much), for a total score ranging from 0 to 28. The ISI was recently validated in a large, heterogeneous sample of cancer patients (Savard, Savard, Simard, & Ivers, 2005).

SECONDARY OUTCOMES:
Modified Edmonton Symptom Assessment System-Revised (ESAS-R) (Philip, Smith, Craft, & Lickiss, (1998) | October 2016 - October 2019, up to 3 years
  A daily assessment of potential side-effects. The ESAS-R assesses symptoms including pain, tiredness, drowsiness, nausea, appetite, shortness of breath, depression, anxiety, and wellbeing on a 0-10 scale. The 9-item measure created for this study includes the pain, drowsiness, depression, anxiety, and wellbeing items and adds fatigue, irritability, forgetfulness, and concentration in a format that otherwise resembles the ESAS-R.
Sleep diary (Carney et al., 2012) | October 2016 - October 2019, up to 3 years
  A standardized daily outcome measure in insomnia research. Each morning respondents require 2-4 minutes to record a) the number of hours slept, b) time in bed, c) sleep onset latency (estimated time in minutes that it took to fall asleep after going to bed), and d) number of awakenings. All medications taken are also recorded. Diary data are used to calculate wake time after sleep onset (the amount of time in bed minus total sleep time and sleep onset latency) and sleep efficiency (the ratio of total sleep time to time in bed).
Positive and Negative Affect Schedule (negative subscale)(Watson, Clark & Tellegen, 1988) | October 2016 - October 2019, up to 3 years
  Comprises of 10 negative adjectives describing emotional states. Using a 5-point scale, respondents rate the extent to which each adjective is consistent with his or her current emotional state.
Pain Intensity Ratings (Jensen, Turner, Romano, & Fisher, 1999) | October 2016 - October 2019, up to 3 years
  Self-reported current, worse, least, and average pain are each assessed. Good validity, reliability, sensitivity to change, and appropriateness to cancer pain have been reported (Jensen et al., 1999).
Functional Assessment of Cancer Therapy-Cognition scale: Perceived Cognitive Impairment subscale (Wagner et al., 2004) | October 2016 - October 2019, up to 3 years
Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS-10) (Espie, Inglis, Harvey, & Tessier, 2000) | October 2016 - October 2019, up to 3 years
  a 10-item self-report measure of maladaptive beliefs about sleep (e.g., beliefs about the immediate and long term negative consequences of insomnia, beliefs about the need for control over insomnia). Although developed as an analogue scale, it was transformed into a Likert-type scale with responses ranging from 1 (strongly disagree) to 6 (strongly agree). Thus, possible scores ranged from 10 to 60, with higher scores indicating more maladaptive cognitions regarding sleep. The DBAS has moderate reliability and validity (Edinger, Wohlegemuth, Radtke, Marsh, & Quillian, 2001).
Pre-Sleep Arousal Scale (PSAS) (Nicassio, Mendlowitz, Fussell, & Petras, 1985) | October 2016 - October 2019, up to 3 years
  An 8-item measure of cognitive hyperarousal associated with insomnia. The subscale score can range from 8 to 40, with higher scores indicating more hyperarousal. Evidence of the internal consistency, test-retest reliability, and convergent validity have been reported by the authors in their initial publication.
Multi-Dimensional Fatigue Inventory (MFI) (Smets, Garssen, Bonke, & de Haes, 1995) | October 2016 - October 2019, up to 3 years
  It consists of 5 subscales, and the authors recommend using the general fatigue subscale for investigations of overall levels of fatigue. The general fatigue (GF) subscale has been found to have good internal consistency (ranging from 0.83-0.90), and GF subscale scores have been shown to positively and significantly correlate with other self-report measures of fatigue. Scores on the sub¬scale range from 4 to 20, with higher scores indicating greater fatigue. It is frequently used with cancer patients (Smets, Garssen, Cull, & de Haes, 1996).
Depression Anxiety Stress Scale - (DASS) (Lovibond & Lovibond, 1995) | October 2016 - October 2019, up to 3 years
  A 42-item self-report measure that can be reliably grouped into three scales: anxiety, depression, and stress; however, only the depression subscale will be included for the present study. The depression subscale has demonstrated high internal consistency (Cronbach's alpha = 0.96) in a clinical sample (Brown, Chorpita, Korotitsch, & Barlow, 1997).
Work and Social Adjustment Scale (WSAS) (Mundt, Marks, Shear, & Griest, 2002) | October 2016 - October 2019, up to 3 years
  A brief, 5-item scale assesses patient's perspectives of impaired functioning in important life domains. The authors report a high level of internal consistency (Cronbach's alpha = .7-.94), good test-retest reliability and sensitivity to change with treatment. Subsequent studies have confirmed its psychometric properties (Mataix-Cols et al., 2006).
Impact of Event Scale (IES) (Horowitz, Wilner, & Alvarez, 1979) | October 2016 - October 2019, up to 3 years
  A 15 item measure of subjective stress in relation to a specific stressor (e.g., cancer). It has strong psychometric properties and is frequently used in cancer research (Cella & Tross, 1986; Cella, Mahon, & Donovan, 1990; Thewes, Meiser, & Hickie, 2001). The four-point frequency scale is as follows: 0='not at all', 1='rarely', 3='sometimes', 5='often', allowing the calculation of a total score (with a possible range of 0-75) and separate intrusion and avoidance subscales scores (with a possible range of 0-35 and 0-40, respectively). Research in oncology suggests a score of ≥ 40 is indicative of a significant stress response (Cella, Mahon, & Donovan, 1990).
Assessment of Survivor Concerns (ASC) (Gotay & Pagano, 2007) | October 2016 - October 2019, up to 3 years
  A 5 item questionnaire designed to measure cancer specific concerns not covered in general quality of life measures. Each item is rated using a four-point Likert scale ranging from 1 (not at all) to 4 (very much). The first three questions load on a cancer-specific worry subscale and the last two measure general health worry. Evidence of internal consistency, convergent and discriminant validity have been demonstrated in the original article. A recent intervention study provides some evidence of its sensitivity to change (Hershman et. al., 2013).
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)- Global Quality of Life Subscale (Aaronson, Ahmedzai, & Bergman, 1993; Osoba et al., 1997) | October 2016 - October 2019, up to 3 years
  Global Quality of Life Subscale (Aaronson, Ahmedzai, & Bergman, 1993; Osoba et al., 1997) was developed and validated with cancer patients. The global quality-of-life scale, comprised of two items rated on a Likert-type scale with responses ranging from 1 (very poor) to 7 (excellent) will be used. Scores are transformed to provide a rating ranging from 0 to 100.
Multi-Dimensional Fatigue Inventory (Smets, Garssen, Bonke, & de Haes, 1995) | October 2016 - October 2019, up to 3 years
Global Adherence Scale | October 2016 - October 2019, up to 3 years
  With acceptable internal consistency (Cronbach's alpha = .81) and construct validity, a modified version of the five-item Medical Outcomes Study General Adherence Scale (MOS-A; Kravitz et al., 1993) assesses compliance with treatment. The MOS-A was modified by replacing physician with psychologist, and sample items are "I followed my psychologist's suggestions exactly" and "I found it easy to do the things my psychologist suggested I do." Participants respond on a scale of 1 (none of the time) to 6 (all of the time). Total scores range from 5 to 30, with higher scores reflecting greater adherence. Scores on the MOS-A have been found to correlate with adherence to other types of regimes in areas of exercise and diet (DiMatteo et al., 1993), and to negatively correlate with barriers to treatment in the area of insomnia (Vincent, Lewycky, & Finnegan, 2008).
Client Feedback Questionnaire | October 2016 - October 2019, up to 3 years
  A four item questionnaire to assess how confident participants are that the online program helped their sleep problem, if they plan to ask for further help (e.g., in person counseling), what they liked best about the program and what they would change to make the program better.
Client Global Improvement and Overall Change (CGI)(Guy, 1976) | October 2016 - October 2019, up to 3 years
  Assesses patients' perceived global improvement. The CGI asked patients to report the overall change in their sleep and in sleep-related effects as a result of participation in their treatment. Participants are asked to rate the change in their sleep and not in any other problem such as chronic pain, depression, or anxiety. Response choices rang from very much improved (1) to very much worse (7). Evidence of the construct validity of the CGI-self-report version comes from the demonstration that CGI scores are significantly and positively associated with treatment-related changes in sleep parameters (e.g., TST, SE) (Vincent, unpublished).

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Harris, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811